CLINICAL TRIAL: NCT00005823
Title: A Randomized Trial for Patients With Acute Myeloid Leukemia or High Risk Myelodysplatic Syndrome Aged 60 or Over
Brief Title: Intensive Compared With Nonintensive Chemotherapy in Treating Older Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leukemia Research Fund (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067831; LRF-AML14; EU-20016; ISRCTN62207270
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2006-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; adult acute monocytic leukemia (M5b); secondary myelodysplastic syndromes; adult acute minimally differentiated myeloid leukemia (M0); atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Cytarabine; Daunorubicin; Etoposide; Hydroxyurea; Idarubicin; Mitoxantrone; Thioguanine; Tretinoin; valspodar

INTERVENTIONS:
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: hydroxyurea
Drug: idarubicin
Drug: mitoxantrone hydrochloride
Drug: thioguanine
Drug: tretinoin
Drug: valspodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known if stronger doses of chemotherapy given over a longer period of time are as well tolerated or as effective as less intensive chemotherapy.

PURPOSE: This randomized phase III trial is studying intensive regimens of chemotherapy to see how well they work compared to nonintensive regimens of chemotherapy in treating older patients with acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate, survival, quality of life, and supportive care requirements with intensive versus nonintensive chemotherapy in older patients with acute myeloid leukemia or high risk myelodysplastic syndrome.
* Compare response achievement, response duration, survival, toxicity and supportive care requirements with differing doses of daunorubicin and cytarabine in these patients receiving intensive chemotherapy.
* Determine the efficacy of PSC 833 in enhancing the effects of daunorubicin in these patients receiving intensive chemotherapy.
* Compare relapse rate, deaths in complete remission, disease free survival, and survival with short versus long intensive chemotherapy in these patients.
* Compare response achievement, response duration, survival, toxicity, quality of life, and resource use with hydroxyurea versus cytarabine in these patients receiving low dose chemotherapy.
* Determine response achievement, response duration, survival, toxicity, quality of life, and supportive care requirements with the addition of tretinoin to the nonintensive chemotherapy in these patients.
* Assess the correlation between P-gp and BCL-2 in family members and treatment outcomes and other prognostic factors in these patients with these treatment regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized or electively assigned to either intensive or nonintensive chemotherapy*.

Intensive chemotherapy

* Induction therapy: Patients are randomized to 1 of 6 treatment arms. Patients receive 2 courses of chemotherapy comprising 1 of 2 daunorubicin doses, 1 of 2 cytarabine doses, thioguanine, and with or without PSC 833.

Patients receive daunorubicin IV once daily on days 1-3 with cytarabine IV twice daily and oral thioguanine once daily on days 1-10 during course 1. Treatment repeats in approximately 31 days as in course 1 except cytarabine and thioguanine are given only on days 1-8.

* Arm I: Patients receive higher dose of daunorubicin, lower dose of cytarabine, and thioguanine.
* Arm II: Patients receive higher dose of daunorubicin, higher dose of cytarabine, and thioguanine.
* Arm III: Patients receive lower dose of daunorubicin, lower dose of cytarabine, and thioguanine.
* Arm IV: Patients receive lower dose of daunorubicin, higher dose of cytarabine, and thioguanine.
* Arm V: Patients receive treatment as in arm III in combination with continuous infusion of PSC 833 beginning day 1.
* Arm VI: Patients receive treatment as in arm IV in combination with continuous infusion of PSC 833 beginning on day 1.

Patients with refractory disease after the first course of induction chemotherapy may continue with the intensive protocol arm or enter the nonintensive arm*. Patients who do not achieve complete remission after completion of induction chemotherapy are removed from study. Patients in complete remission after induction therapy receive consolidation therapy.

* Consolidation therapy: Patients in complete remission after induction are randomized to either short or long consolidation.

  * Short consolidation: Patients receive mitoxantrone IV on days 1-3 and cytarabine IV over 2 hours twice daily on days 1-3.
  * Long consolidation: Patients complete short consolidation and then receive idarubicin IV over 5 minutes once daily on days 1 and 3, cytarabine IV over 2 hours twice daily and etoposide IV over 1 hour once daily on days 1-3.

Non-intensive chemotherapy*

* Patients are randomized to 1 of 4 treatment arms.

  * Arm I: Patients receive oral hydroxyurea as necessary to control WBC count until treatment failure.
  * Arm II: Patients receive hydroxyurea as in arm I and oral tretinoin daily for up to 16 weeks.
  * Arm III: Patients receive low dose cytarabine subcutaneously twice daily on days 1-10 every 28 days for a minimum of 4 courses.
  * Arm IV: Patients receive cytarabine as in arm III plus oral tretinoin daily for up to 16 weeks.

NOTE: *Patients with liver function test > 2 times upper limit of normal are not eligible for nonintensive randomization

Quality of life is assessed at study entry, and then at 1, 3, and 6 months.

Patients are followed at one year.

PROJECTED ACCRUAL: Approximately 2,000 patients (1,200 to intensive arm and 800 to nonintensive arm) will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Acute myeloid leukemia (de novo or secondary) OR
* Myelodysplastic syndrome

  * More than 10% myeloblasts in the bone marrow
  * Refractory anemia with excess blasts
  * Refractory anemia with excess blasts in transformation
  * Chronic myelomonocytic leukemia
* No acute promyelocytic leukemia (FAB type M3)
* No blastic phase chronic myeloid leukemia

PATIENT CHARACTERISTICS:

Age:

* 60 and over (younger patients allowed if intensive chemotherapy not indicated)

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No liver function test ≥ 2 times normal (for non-intensive therapy arm)

Renal:

* Not specified

Cardiovascular:

* No myocardial infarction within past 6 months in patients receiving daunorubicin or PSC 833

Other:

* No other concurrent active malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy for leukemia

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 1998-12; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Survival
Response achievement
Response duration

SECONDARY OUTCOMES:
Toxicity by WHO Toxicity Grading after each treatment course
Quality of life EORTC QLQ-C30 at 3 days, 1 month, 3 months, and 6 months from study entry
Resource use (use of blood products, antibiotics and days in hospital) after each treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Alan K. Burnett, MD, FRCP, Study Chair — University Hospital of Wales
Locations (3):
- United Kingdom (3):
  - Queen Elizabeth Hospital at University of Birmingham, Birmingham, England
  - University College Hospital, London, England
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Background] Seedhouse CH, Grundy M, White P, Li Y, Fisher J, Yakunina D, Moorman AV, Hoy T, Russell N, Burnett A, Pallis M; National Cancer Research Network. Sequential influences of leukemia-specific and genetic factors on p-glycoprotein expression in blasts from 817 patients entered into the National Cancer Research Network acute myeloid leukemia 14 and 15 trials. Clin Cancer Res. 2007 Dec 1;13(23):7059-66. doi: 10.1158/1078-0432.CCR-07-1484. PMID 18056183
- [Background] Burnett AK, Milligan D, Hills RK, et al.: Does all-transretinoic acid (ATRA) have a role in non-APL acute myeloid leukaemia? Results from 1666 patients in three MRC trials. [Abstract] Blood 104 (11): A-1794, 2004.
- [Result] Burnett AK, Milligan D, Goldstone A, Prentice A, McMullin MF, Dennis M, Sellwood E, Pallis M, Russell N, Hills RK, Wheatley K; United Kingdom National Cancer Research Institute Haematological Oncology Study Group. The impact of dose escalation and resistance modulation in older patients with acute myeloid leukaemia and high risk myelodysplastic syndrome: the results of the LRF AML14 trial. Br J Haematol. 2009 May;145(3):318-32. doi: 10.1111/j.1365-2141.2009.07604.x. Epub 2009 Mar 8. PMID 19291085
- [Result] Burnett AK, Milligan D, Prentice AG, Goldstone AH, McMullin MF, Hills RK, Wheatley K. A comparison of low-dose cytarabine and hydroxyurea with or without all-trans retinoic acid for acute myeloid leukemia and high-risk myelodysplastic syndrome in patients not considered fit for intensive treatment. Cancer. 2007 Mar 15;109(6):1114-24. doi: 10.1002/cncr.22496. PMID 17315155
- [Result] Burnett AK, Milligan DW, Prentice AG, et al.: Modification or dose or treatment duration has no impact on outcome of AML in older patients: preliminary results of the UK NCRI AML14 trial. [Abstract] Blood 106 (11): A-543, 2005.
- [Result] Burnett AK, Milligan D, Prentice AG, et al.: Low dose Ara-C versus hydroxyurea with or without retinoid in older patients not considered fit for intensive chemotherapy: the UK NCRI AML14 trial. [Abstract] Blood 104 (11): A-872, 2004.
- [Result] Pallis M, Truran L, Grundy M, et al.: P-Glycoprotein overexpresion and internal tandem duplications of FLT3 are characteristic of discrete populations of elderly AML patients. [Abstract] Blood 104 (11): A-196, 2004.